CLINICAL TRIAL: NCT04212949
Title: The Effect of Transcranial Magnetic Stimulation Therapy Combined With Transforaminal Epidural Steroid Injection in Patients With Lumbar Radiculopathy
Brief Title: The Effect of Transcranial Magnetic Stimulation Therapy in Patients With Lumbar Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2019.983
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Lumbar Radiculopathy
Keywords: lumbar radiculopathy; rTMS; TESI; treatment
MeSH Terms: conditions — Radiculopathy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive transcranial magnetic stimulation following TESI (Experimental): Active repetitive transcranial magnetic stimulation will be performed to the patients with lumbar radiculopathy who receive transforaminal epidural steroid injection.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS); Drug: Transforaminal epidural steroid injection
- Transforaminal epidural steroid injection (Active Comparator): Transforaminal epidural steroid injection will be applied to the patients with lumbar radiculopathy.
  Interventions: Drug: Transforaminal epidural steroid injection

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — Stimulation will be performed from the contralateral M1 cortex of the painful side. Each stimulation session will consist of 1500 pulses (30 trains of 5 seconds each, with an inter-train interval of 25 seconds) delivered at a frequency of 10 Hz. The stimulation intensity will be set at 80% of the resting motor threshold.
  Arms: Repetitive transcranial magnetic stimulation following TESI
Drug: Transforaminal epidural steroid injection — An epidural steroid injection under guidance of fluoroscopy is used to reduce inflammation at a lumbar spinal nerve root(s).
  The following drugs will be used for this procedure: 80mg/2ml triamcinolone acetonide (sinakort-A) and 1 mL 0.5% bupivacaine (marcaine)

SUMMARY:
The present study aims to investigate the efficacy of repetitive transcranial magnetic stimulation of the motor cortex combined with transforaminal epidural steroid injection in patients with chronic lumbar radiculopathy.

DETAILED DESCRIPTION:
Treatment methods of lumbar radiculopathy include short-term bed rest, medical treatments, physical therapy and rehabilitation techniques, psychotherapy, acupuncture, cryotherapy, epidural steroid injections, and surgical treatment. Epidural steroid injection is an effective treatment procedure in patients whose conservative treatment methods are not successful. Fluoroscopy guided transforaminal epidural steroid injection (TESI) is the most ideal procedure and it is considered as an effective treatment approach in radicular pain and concomitant neuropathic pain because of reaching the target area, which is the origin of pathology. Although radicular pain is usually caused by a peripheral lesion, central sensitization and maladaptive plasticity have been shown to play an important role in the development and chronicity of this pain. These data suggest that central pain processing should be altered or stopped, especially in the presence of refractory pain. Repetitive transcranial magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS) are non-invasive brain stimulation techniques that are increasingly being used to treat refractory neuropathic pain. Although short-term efficacy of rTMS treatment in radicular pain management was shown in one study, long-term efficacy was not evaluated and the necessity of trials evaluating long-term efficacy was reported. In accordance with these findings, we aimed to investigate the long-term effect of rTMS treatment in patients with chronic lumbar radiculopathy who received TESI.

Patients diagnosed with chronic lumbar radiculopathy and planned to administer fluoroscopy-guided TESI will be included in the study. Patients will be randomized into two groups following TESI. Home-based exercise program will be given to both groups after injection. One week after the injection, only the first group will receive 10 sessions of rTMS treatment for 2 weeks in addition to the exercise program. rTMS treatment will be performed with the device used in our clinic for neurological rehabilitation and pain management.

Patients will be assessed by a blind researcher using the Visual Analogue Scale (VAS) for low back and leg pain, the Douleur Neuropathique 4 Questions (DN-4) for neuropathic pain, the Oswestry Disability Index for disability, the Beck Depression Scale for depression, and the Central Sensitization Inventory for central sensitization. All assessments will be performed by the same physician before injection, first hour (only VAS), third week, third month, and sixth month after the injection. All adverse events will be noted.

After data collection, analysis will be performed with the appropriate statistical method.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 20-60 years
2. Symptoms lasting longer than 3 months
3. To be planned TESI due to root compression which is caused by lumbar disk herniation
4. To agree to participate in the study

Exclusion Criteria:

1. Lumbar spinal stenosis
2. Presence of clinical findings incompatible with MRI
3. Spinal disease (trauma / tumor)
4. Spondylodiscitis or inflammatory spondylitis
5. Presence of epilepsy
6. Presence of implanted medical devices such as pacemakers, insulin pumps
7. Intracranial metallic implant
8. Previous cranial surgery history
9. Brain tumor
10. Severe hearing and vision loss
11. To be applied TESI for the last six months
12. Presence of surgical history through lumbar region
13. Scoliosis
14. Spodilolistezis
15. Pregnancy
16. Osteoporotic lumbar fracture
17. The presence of inflammatory diseases that affect spinal morphology, such as ankylosing spondylitis
18. Patients with electrophysiologically determined polyneuropathy, amyotrophic lateral sclerosis, etc. neurological disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-11-08 (Estimated); Study Completion 2020-12-08 (Estimated)

PRIMARY OUTCOMES:
Low back and leg pain | before treatment (T0)
  Low back and leg pain will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no pain) to "10 cm" (intolerable pain).
Low back and leg pain | 1st hour after injection (T1)
  Low back and leg pain will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no pain) to "10 cm" (intolerable pain).
Low back and leg pain | 3rd week of treatment (T2)
  Low back and leg pain will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no pain) to "10 cm" (intolerable pain).
Low back and leg pain | 3rd month of treatment (T3)
  Low back and leg pain will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no pain) to "10 cm" (intolerable pain).
Low back and leg pain | 6th month of treatment (T4)
  Low back and leg pain will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no pain) to "10 cm" (intolerable pain).

SECONDARY OUTCOMES:
Quality of life and activities of daily living | before treatment (T0)
  The potential changes in quality of life and activities of daily living will be measured by validated Oswestry Disability Index scores. It consists of 10 questions and the patient gets a minimum of "0" and a maximum of "5" points for each question. According to this, it is calculated how many percent of the patient's life activities are affected. Higher scores mean a worse outcome.
Quality of life and activities of daily living | 3rd week of treatment (T1)
  The potential changes in quality of life and activities of daily living will be measured by validated Oswestry Disability Index scores. It consists of 10 questions and the patient gets a minimum of "0" and a maximum of "5" points for each question. According to this, it is calculated how many percent of the patient's life activities are affected. Higher scores mean a worse outcome.
Quality of life and activities of daily living | 3rd month of treatment (T2)
  The potential changes in quality of life and activities of daily living will be measured by validated Oswestry Disability Index scores. It consists of 10 questions and the patient gets a minimum of "0" and a maximum of "5" points for each question. According to this, it is calculated how many percent of the patient's life activities are affected. Higher scores mean a worse outcome.
Quality of life and activities of daily living | 6th month of treatment (T3)
  The potential changes in quality of life and activities of daily living will be measured by validated Oswestry Disability Index scores. It consists of 10 questions and the patient gets a minimum of "0" and a maximum of "5" points for each question. According to this, it is calculated how many percent of the patient's life activities are affected. Higher scores mean a worse outcome.
Neuropathic pain | before treatment (T0)
  Douleur Neuropathique 4 questions will be used to determine the presence of neuropathic pain. It consists of ten questions, 7 questions are related with symptoms and the answer to the other 3 questions is determined by clinical examination. Scoring is between 0 and10 and a score of 4 and above is considered as neuropathic pain.
Neuropathic pain | 3rd week of treatment (T1)
  Douleur Neuropathique 4 questions will be used to determine the presence of neuropathic pain. It consists of ten questions, 7 questions are related with symptoms and the answer to the other 3 questions is determined by clinical examination. Scoring is between 0 and10 and a score of 4 and above is considered as neuropathic pain.
Neuropathic pain | 3rd month of treatment (T2)
  Douleur Neuropathique 4 questions will be used to determine the presence of neuropathic pain. It consists of ten questions, 7 questions are related with symptoms and the answer to the other 3 questions is determined by clinical examination. Scoring is between 0 and10 and a score of 4 and above is considered as neuropathic pain.
Neuropathic pain | 6th month of treatment (T3)
  Douleur Neuropathique 4 questions will be used to determine the presence of neuropathic pain. It consists of ten questions, 7 questions are related with symptoms and the answer to the other 3 questions is determined by clinical examination. Scoring is between 0 and10 and a score of 4 and above is considered as neuropathic pain.
Central sensitization | before treatment (T0)
  Central sensatization inventory will be used to identify the presence and severity of central sensitization. Central Sensatization Inventory consists of 25 questions. Each question is scored between 0 and 4 (0 = never, 4 = always). A score of 40 or above indicates the presence of central sensitization with 81% sensitivity and 75% specificity. Central sensitization severity was defined as 0-29 subclinical, 30-39 mild, 40-49 moderate, 50-59 severe, >59 very severe. Higher scores mean a worse outcome.
Central sensitization | 3rd week of treatment (T1)
  Central sensatization inventory will be used to identify the presence and severity of central sensitization. Central Sensatization Inventory consists of 25 questions. Each question is scored between 0 and 4 (0 = never, 4 = always). A score of 40 or above indicates the presence of central sensitization with 81% sensitivity and 75% specificity. Central sensitization severity was defined as 0-29 subclinical, 30-39 mild, 40-49 moderate, 50-59 severe, >59 very severe. Higher scores mean a worse outcome.
Central sensitization | 3rd month of treatment (T2)
  Central sensatization inventory will be used to identify the presence and severity of central sensitization. Central Sensatization Inventory consists of 25 questions. Each question is scored between 0 and 4 (0 = never, 4 = always). A score of 40 or above indicates the presence of central sensitization with 81% sensitivity and 75% specificity. Central sensitization severity was defined as 0-29 subclinical, 30-39 mild, 40-49 moderate, 50-59 severe, >59 very severe. Higher scores mean a worse outcome.
Central sensitization | 6th month of treatment (T3)
  Central sensatization inventory will be used to identify the presence and severity of central sensitization. Central Sensatization Inventory consists of 25 questions. Each question is scored between 0 and 4 (0 = never, 4 = always). A score of 40 or above indicates the presence of central sensitization with 81% sensitivity and 75% specificity. Central sensitization severity was defined as 0-29 subclinical, 30-39 mild, 40-49 moderate, 50-59 severe, >59 very severe. Higher scores mean a worse outcome.
The Beck depression inventory | before treatment (T0)
  The Beck depression inventory is a 21-item, self-rated scale that evaluates key symptoms of depression including mood, pessimism, sense of failure, self-dissatisfaction, guilt, punishment, self-dislike, self-accusation, suicidal ideas, crying, irritability, social withdrawal, indecisiveness, body image change, work difficulty, insomnia, fatigability, loss of appetite, weight loss, somatic preoccupation, and loss of libido. The minimum score is 0 and the maximum score is 63. Higher scores mean a worse outcome. Higher scores indicate the severity of depression.
The Beck depression inventory | 3rd week of treatment (T1)
  The Beck depression inventory is a 21-item, self-rated scale that evaluates key symptoms of depression including mood, pessimism, sense of failure, self-dissatisfaction, guilt, punishment, self-dislike, self-accusation, suicidal ideas, crying, irritability, social withdrawal, indecisiveness, body image change, work difficulty, insomnia, fatigability, loss of appetite, weight loss, somatic preoccupation, and loss of libido. The minimum score is 0 and the maximum score is 63. Higher scores mean a worse outcome. Higher scores indicate the severity of depression.
The Beck depression inventory | 3rd month of treatment (T2)
  The Beck depression inventory is a 21-item, self-rated scale that evaluates key symptoms of depression including mood, pessimism, sense of failure, self-dissatisfaction, guilt, punishment, self-dislike, self-accusation, suicidal ideas, crying, irritability, social withdrawal, indecisiveness, body image change, work difficulty, insomnia, fatigability, loss of appetite, weight loss, somatic preoccupation, and loss of libido. The minimum score is 0 and the maximum score is 63. Higher scores mean a worse outcome. Higher scores indicate the severity of depression.
The Beck depression inventory | 6th month of treatment (T3)
  The Beck depression inventory is a 21-item, self-rated scale that evaluates key symptoms of depression including mood, pessimism, sense of failure, self-dissatisfaction, guilt, punishment, self-dislike, self-accusation, suicidal ideas, crying, irritability, social withdrawal, indecisiveness, body image change, work difficulty, insomnia, fatigability, loss of appetite, weight loss, somatic preoccupation, and loss of libido. The minimum score is 0 and the maximum score is 63. Higher scores mean a worse outcome. Higher scores indicate the severity of depression.
Adverse events | before treatment (T0)
  All adverse events and complications will be noted.
Adverse events | 1st hour after injection (T1)
  All adverse events and complications will be noted.
Adverse events | 3rd week of treatment (T2)
  All adverse events and complications will be noted.
Adverse events | 3rd month of treatment (T3)
  All adverse events and complications will be noted.
Adverse events | 6th month of treatment (T4)
  All adverse events and complications will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gündüz, Prof, Study Chair — Marmara University; Gülseren Akyüz, Prof, Study Chair — Marmara University
Locations (1):
- Marmara University School of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang SS, Hwang BM, Son HJ, Cheong IY, Lee SJ, Lee SH, Chung TY. The dosages of corticosteroid in transforaminal epidural steroid injections for lumbar radicular pain due to a herniated disc. Pain Physician. 2011 Jul-Aug;14(4):361-70. PMID 21785479
- [Background] Attal N, Ayache SS, Ciampi De Andrade D, Mhalla A, Baudic S, Jazat F, Ahdab R, Neves DO, Sorel M, Lefaucheur JP, Bouhassira D. Repetitive transcranial magnetic stimulation and transcranial direct-current stimulation in neuropathic pain due to radiculopathy: a randomized sham-controlled comparative study. Pain. 2016 Jun;157(6):1224-1231. doi: 10.1097/j.pain.0000000000000510. PMID 26845524
- [Background] Roussel NA, Nijs J, Meeus M, Mylius V, Fayt C, Oostendorp R. Central sensitization and altered central pain processing in chronic low back pain: fact or myth? Clin J Pain. 2013 Jul;29(7):625-38. doi: 10.1097/AJP.0b013e31826f9a71. PMID 23739534
- [Background] Galhardoni R, Correia GS, Araujo H, Yeng LT, Fernandes DT, Kaziyama HH, Marcolin MA, Bouhassira D, Teixeira MJ, de Andrade DC. Repetitive transcranial magnetic stimulation in chronic pain: a review of the literature. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S156-72. doi: 10.1016/j.apmr.2014.11.010. Epub 2014 Nov 28. PMID 25437106
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Sari S, Aydin ON, Guleser G, Kurt I, Turan A. Effect of transforaminal anterior epidural steroid injection on neuropathic pain, quality of sleep and life. Agri. 2015;27(2):83-8. doi: 10.5505/agri.2015.91489. PMID 25944134